CLINICAL TRIAL: NCT07359352
Title: Surgical Care And Recovery With Laser Evaluation Trial (SCARLET)
Acronym: SCARLET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2379205
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Post-surgical Scars; Hypertrophic Scars; Scar Appearance Dissatisfaction; Aesthetic Surgical Outcomes; Wound Healing After Body-contouring Surgery
Keywords: Surgical scar; Postoperative scar; Hypertrophic scar; Body-contouring surgery; Abdominoplasty scar; Brachioplasty scar; Thighplasty scar; Scar revision; Laser-assisted scar remodeling
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a prospective, two-arm, parallel-group, single-center cohort study comparing postoperative scar outcomes between:
  Cosmetic Group - receiving three sessions of ProFractional laser and/or Broadband Light (BBL) therapy at approximately 4, 8, and 14 weeks postoperatively, and
  Non-Cosmetic Group - receiving standard postoperative care only. Both groups complete standardized scar assessments (SCAR-Q, POSAS) and undergo photographic documentation at predefined intervals up to 6 months after surgery.
Who Masked: Outcomes Assessor
Masking Description: Participants and providers are aware of treatment allocation; however, photographic scar evaluations are conducted by blinded assessors who do not have access to participant group assignments or treatment histories. This ensures objectivity in evaluating visual scar outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cosmetic Group (Laser/BBL Therapy) (Experimental): Participants in this group will receive three sessions of ProFractional laser and/or Broadband Light (BBL) therapy following their qualifying body-contouring surgical procedure. Treatments will begin approximately 4 weeks postoperatively, with subsequent sessions at 8 weeks and 14 weeks (±2 weeks).
  Laser parameters will be determined by the treating provider based on clinical assessment and Fitzpatrick Skin Type.
  Assessments will include standardized scar photographs, SCAR-Q, and POSAS questionnaires at each visit and at 6 months postoperatively.
  The objective is to determine whether early adjuvant energy-based therapy improves scar quality, appearance, and patient-reported satisfaction compared to standard care.
  Interventions: Device: ProFractional Laser Therapy and/or Broadband Light (BBL) Treatment
- Non-Cosmetic Group (Standard Postoperative Care) (No Intervention): Participants in this group will undergo standard postoperative wound management without laser or BBL therapy.
  They will complete the same follow-up visits and outcome assessments as the cosmetic group-including SCAR-Q and POSAS questionnaires, and standardized photographic documentation-at 4, 8, and 14 weeks, and 6 months postoperatively.
  This group serves as a comparator to evaluate the natural progression of scar healing and satisfaction under standard care conditions.

INTERVENTIONS:
Device: ProFractional Laser Therapy and/or Broadband Light (BBL) Treatment — ProFractional laser creates microthermal injury zones that stimulate collagen remodeling and accelerate re-epithelialization.
  Broadband Light (BBL) therapy uses filtered pulsed light to target hemoglobin and melanin, reducing erythema and pigmentation while promoting dermal repair.
  Each participant in the cosmetic arm will receive up to three sessions spaced 4-6 weeks apart, using device settings individualized by the investigator to the participant's scar characteristics and skin type.
  All treatments are performed by trained and credentialed clinical staff in accordance with manufacturer safety guidelines and AdventHealth institutional standards.
  Arms: Cosmetic Group (Laser/BBL Therapy)

SUMMARY:
The Surgical Care and Recovery with Laser Evaluation Trial (S.C.A.R.L.E.T.) is a prospective, single-center clinical study conducted at AdventHealth Medical Group Plastic and Reconstructive Surgery at Innovation Tower. The study evaluates whether early adjuvant ProFractional laser and/or Broadband Light (BBL) therapy improves the appearance, texture, and patient-reported outcomes of surgical scars following major body-contouring procedures. Participants undergoing qualifying surgeries will be grouped as either cosmetic (receiving three laser/BBL sessions) or non-cosmetic (receiving standard care only). Scar outcomes will be assessed using validated instruments-SCAR-Q and Patient and Observer Scar Assessment Scale (POSAS)-along with standardized photographic analysis at serial follow-ups through six months postoperatively.

DETAILED DESCRIPTION:
Surgical body-contouring procedures often produce long, visible scars that can affect patient satisfaction and quality of life. This study aims to determine whether early initiation of fractional laser or BBL therapy can enhance wound remodeling, reduce scar revision rates, and improve overall aesthetic and psychosocial outcomes compared to standard postoperative care.

Eligible adult participants (≥18 years) scheduled for body-contouring procedures-including brachioplasty, chest/breast contouring, abdominoplasty/panniculectomy, buttock/lower-body lift, or thighplasty-will be enrolled. Participants will be assigned to one of two cohorts:

Cosmetic Group: Will receive three sessions of laser and/or BBL therapy at approximately 4, 8, and 14 weeks postoperatively, following established safety parameters.

Non-Cosmetic Group: Will receive standard postoperative care without adjuvant light-based treatment.

Both groups will complete the SCAR-Q and POSAS questionnaires at 4, 8, 14 weeks, and 6 months after surgery. Standardized photographs of the surgical site will be taken at each visit for blinded evaluation of scar color, texture, and overall quality. Fitzpatrick Skin Type will be recorded for subgroup analysis.

The primary objective is to determine whether early adjuvant laser/BBL therapy produces statistically significant and clinically meaningful improvements in scar quality-based on SCAR-Q and POSAS scores-compared to standard care.

The secondary objective is to assess whether adjuvant treatment reduces the incidence of surgical scar revisions within the first postoperative year.

The study will enroll approximately 150 participants and is expected to take up to 24 months for recruitment with a total study duration of 36 months (including analysis). Statistical analyses will include repeated measures ANOVA and Chi-square tests with α = 0.05.

Safety assessments will include documentation of adverse events related to both surgery and light-based therapy (e.g., erythema, hyperpigmentation, infection, or delayed wound healing). All laser treatments will be performed by qualified providers in accordance with manufacturer guidelines and institutional protocols.

No compensation is provided to participants. Findings are intended for publication in peer-reviewed surgical or aesthetic medicine journals to improve evidence-based postoperative scar management strategies.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older.

Scheduled to undergo one or more of the following major body-contouring procedures during the study period:

Brachioplasty (arm lift)

Chest or breast contouring surgery

Abdominoplasty or panniculectomy

Buttock lift or lower body lift

Thighplasty (thigh lift)

Able and willing to provide written informed consent.

Able to read and write in English (required for completion of validated questionnaires).

Willing and able to comply with scheduled follow-up visits, questionnaires, and study procedures for up to 12 months post-surgery.

Exclusion Criteria:

Inability or unwillingness to provide informed consent.

Inability to comply with study visits or procedures.

Non-English speakers, as the validated SCAR-Q and POSAS instruments are not currently available in equivalent translations.

Current use of nicotine or nicotine-containing products, including cigarettes, vaping, chewing tobacco, or nicotine replacement therapy, due to the known adverse effects of nicotine on wound healing and scar formation.

Any medical condition, treatment, or circumstance that, in the opinion of the Investigator, may increase participant risk, compromise safety, or interfere with study participation or data integrity.

Pregnant or breastfeeding women (laser/BBL therapy contraindicated in pregnancy).

History of abnormal scar formation such as keloids or hypertrophic scarring (if deemed clinically significant by the investigator).

Recent energy-based treatment (laser, IPL, or BBL) to the surgical site within the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in SCAR-Q Total Score from Baseline to 6 Months Post-Surgery | Baseline (Preoperative) to 6 months post-surgery (±1 month)
  The SCAR-Q is a validated, patient-reported outcome instrument designed to assess appearance, symptoms (such as pain, itchiness, and tightness), and psychosocial impact of scarring.
  Scores are transformed on a 0-100 scale, with higher scores indicating better scar-related quality of life and aesthetic satisfaction.
  The change in total and domain-specific SCAR-Q scores from baseline to six months postoperatively will be compared between participants receiving ProFractional laser/BBL therapy and those receiving standard postoperative care.

SECONDARY OUTCOMES:
Change in POSAS (Patient and Observer Scar Assessment Scale) Score from Baseline to 6 Months Post-Surgery | Baseline (Preoperative) to 6 months post-surgery (±1 month)
  The POSAS is a hybrid assessment tool composed of patient and observer subscales evaluating scar pigmentation, thickness, surface relief, pliability, pain, and itch.
  Lower scores indicate scars more similar to normal skin. Both patient and observer scores will be collected at each postoperative timepoint and compared longitudinally between intervention and control groups.
Surgical Scar Revision Rate | Baseline (Surgery Day) to 12 months post-surgery
  The proportion of participants requiring surgical scar revision within 12 months postoperatively will be compared between the laser/BBL and standard care groups.
  Scar revision is defined as any re-excision, laser resurfacing, or procedural intervention performed specifically to improve the cosmetic or structural quality of a prior surgical scar.

OTHER OUTCOMES:
Photographic Evaluation of Scar Appearance | 4 weeks, 8 weeks, 14 weeks, and 6 months post-surgery.
  Standardized photographs of surgical sites will be collected at each follow-up visit under controlled lighting and positioning. Blinded evaluators will assess photographs using visual analog scales for pigmentation, surface texture, and overall aesthetic improvement.
Patient Global Satisfaction Rating | 6 months post-surgery.
  Participants will rate their overall satisfaction with scar appearance and comfort on a Likert scale from "Very Dissatisfied" to "Very Satisfied."
Incidence of Adverse Events Related to Scar Management | From first laser/BBL treatment through 6-month follow-up.
  Adverse events such as erythema, hyperpigmentation, infection, or delayed wound healing will be monitored throughout the study and classified by severity and relationship to the intervention.

IPD SHARING:
Plan to Share IPD: Undecided
We will not be sharing information from this study, but will be publishing information in scientific journals.

REFERENCES:
- [Result] Chung JH, Kim DS, Cheon JH, Yoon JM, Baek SK, Jung KY, Yoon ES, Park SH. Current Protocol for Aesthetic Scar Management in Thyroid Surgery. Laryngoscope. 2021 Jul;131(7):E2188-E2195. doi: 10.1002/lary.29441. Epub 2021 Feb 10. PMID 33567135
- [Result] Cohen JL. Minimizing skin cancer surgical scars using ablative fractional Er:YAG laser treatment. J Drugs Dermatol. 2013 Oct;12(10):1171-3. PMID 24085055
- [Result] Tanzi EL, Alster TS. Single-pass carbon dioxide versus multiple-pass Er:YAG laser skin resurfacing: a comparison of postoperative wound healing and side-effect rates. Dermatol Surg. 2003 Jan;29(1):80-4. doi: 10.1046/j.1524-4725.2003.29012.x. PMID 12534517